CLINICAL TRIAL: NCT00490373
Title: A Phase 2 Trial of ALIMTA in Pretreated Patients With Unresectable or Metastatic Cancer of the Pancreas
Brief Title: Trial of Pemetrexed for Patients With Pancreatic Cancer Which Cannot be Treated With Surgery or is Metastatic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8621; H3E-SB-S041
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pemetrexed

SUMMARY:
This study with pemetrexed is for patients with metastatic or unresectable pancreatic cancer who progressed after first line chemotherapy with gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of adenocarcinoma of the pancreas that is locally advanced (Stage II, III) or metastatic (Stage IV), as staged by the American Joint Committee on Cancer (AJCC; Protocol Attachment S041.2; Fleming et al. 1997), and not amenable to resection with curative intent.
* Prior systemic first line chemotherapy with gemcitabine single agent or a combination regimen including gemcitabine (not more than one prior systemic chemotherapy allowed).
* Uni-dimensionally measurable disease according to the RECIST criteria (Therasse et al. 2000), defined as: At least one lesion that can be accurately measured in at least one dimension, with the longest diameter greater than or equal to 2 cm with conventional techniques or greater than or equal to 1.0 cm with spiral CT scans. Ultrasound and X-ray are NOT allowed to measure or follow lesions.

Exclusion Criteria:

* Prior radiation of equal to or greater than 25% of the bone marrow (Cristy and Eckerman 1987)
* Prior immunotherapy, biological therapy, and/or hormonal therapy for pancreas cancer.
* Prior systemic chemotherapy with 5-FU.
* Patient not yet recovered from the acute toxic effects of the treatment prior to study enrollment.
* Radiotherapy within the last 4 weeks before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-10; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy.

SECONDARY OUTCOMES:
To assess tumor response.
To assess time to event efficacy variables including time to progressive disease and overall survival.
To characterize the quantitative and qualitative toxicities of pemetrexed in this population of pancreatic cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt, Germany

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com